CLINICAL TRIAL: NCT00202111
Title: Australasian Multicentered Prospective Randomised Clinical Study Comparing Laparoscopic and Conventional Open Surgical Treatments of Colon Cancer in Adults
Brief Title: Comparative Study of Laparoscopic Versus Open Operations for Colon Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Queen Elizabeth Hospital (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Health Research Council, New Zealand (Other); Ethicon Endo-Surgery (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 83449871; NH&MRC ID 207815; NH&MRC ID 349381
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-10-17 (Estimated); Status verified 2006-02

CONDITIONS: Colonic Neoplasms
Keywords: Clinical Trial; Colonic Neoplasms; Laparoscopic Surgery; Morbidity; Port Site Metastasis; Disease-Free Survival
MeSH Terms: conditions — Colonic Neoplasms

INTERVENTIONS:
Procedure: Laparoscopic-assisted colectomy
Procedure: Conventional open colectomy

SUMMARY:
The purpose of this study is to compare the short and long term outcomes of people who have colon cancers removed either by laparotomy (a large cut in the abdominal wall) or by a laparoscopic assisted approach (keyhole surgery). This study involves 37 credentialled surgeons in 20 approved hospitals across Australasia and during the recruitment period (Jan 1998 to March 2005) 601 patients were recruited into the ALCCaS Trial.

DETAILED DESCRIPTION:
AIMS

The primary aim of the study is to test the hypothesis that tumour related disease free interval and overall survival are equivalent regardless whether patients receive laparoscopic colon resection (LCR) or open colon resection (OCR) at three and five years post operatively. The secondary aims of the study are to determine the safety of LCR compared to OCR and 30 day mortality and compare post operative pain, paralytic ileus, early and late morbidities (including wound site recurrence), recovery, transfusion requirements, cost and quality of life scores.

BACKGROUND

The ALCCaS Trial is an Australasian, multicentred, prospective, randomised clinical study comparing laparoscopic and conventional open surgical treatments of colon cancer in adults. This trial has been recruiting patients since 1998.

Patients are randomised to receive either laparoscopic or conventional open resection for colon cancer. A Randomisation Centre was established to provide a 24-hour randomisation service and this centre is situated in Christchurch, New Zealand. The Health Research Council of New Zealand Data Safety Committee, chaired by Professor Tom Fleming, access the ALCCaS Trial annually to ensure that it meets strict ethical and research related criteria.

During the recruitment period (Jan 1998 to March 2005) 601 patients were recruited into the ALCCaS Trial. There have been 37 surgeons involved in recruiting patients at 20 hospitals within Australia and New Zealand. All surgeons participating in the ALCCaS trial are accredited in laparoscopic surgical techniques. To gain accreditation, a surgeon must have carried out no less than 20 supervised colon resections and must provide video evidence of two laparoscopic colonic resections for review. Surgeons from throughout Australia and New Zealand are participating in this study. The Research Ethics Committees at a variety of hospitals throughout New South Wales, Queensland, South Australia, Victoria, Western Australia and New Zealand have approved the study.

DATA COLLECTION

The type of colon resection performed by the individual surgeon will follow standard oncologically safe principles. The following intra-operative details will be collected, the patient epidemiology, ASA status, previous abdominal surgery, incision type, site of carcinoma, modality of diagnosis, pre operative haemoglobin and lung function tests, pre operative blood transfusion, planned operation, planned incision. Intra operatively the date of the operation, whether DVT prophylaxis has been used, the type of bowel preparation, the type of operation performed, if the laparoscopic procedure is performed whether it included mobilisation of the bowel, ligation of main artery and vein, transection of the bowel, resection of the bowel and anastomosis done as an intraperitoneal procedure are recorded.

The use of cytotoxic irrigation of the peritoneum, wound and colonic lumen is noted. Estimated surgical blood loss and intra operative blood transfusion is recorded. The post operative position of the tumour is noted. The type of incision and size of incision is recorded. Any reason for change in planned incision is recorded and the theatre utilisation, and total anaesthetic time and duration of the operative procedure are recorded. Intra operative temperature record is kept. Reason for stoma formation, if applicable, is recorded. The intra operative costs and disposable items are identified. Intra operative complications are identified as well as adverse events involving surgical equipment.

In the post operative phase the total intravenous fluid requirement, blood transfusion, pain scores, amount of Morphine used, whether the patient vomited and whether nasogastric tube is required as well as lung function tests and any adverse events are noted at 30 minutes following the procedure, 6 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours, 168 hours and continued daily until the patient is discharged if not already discharged at that time. At discharge from hospital, total hospital days are identified as well as time in high dependency unit or intensive care unit, reason for delay in discharge is noted, post operative events including cardiac, respiratory, renal, ileus, wound infection, anastomotic leakage and other events are identified.

Pathology includes the site of tumour, TNM staging, ACPS staging, length of resected colon, proximal clearance, distal clearance, number of nodes obtained, tumour differentiation, venous invasion, perineal invasion and histological type. Adjuvant chemotherapy if planned is noted. Patients in the study may be entered into an adjuvant chemotherapy trial following surgery provided the subsequent trial does not have radiation as a component of therapy and that the chemotherapy trial allows entering of patients from both surgical arms of the study. Follow up is quarterly for the first year, 6 monthly for year two and three and then annually until year five. At follow up wounds are check for any evidence of recurrence. A colonoscopy is performed 12 months following resection and then every three years following that if negative. Chest xray, abdominal CT or liver ultrasound, a complete blood picture are performed if clinically indicated, CEA's performed six monthly.

FOLLOW-UP SCHEDULE

Patients are followed for tumour recurrence and survival. Patients are advised on, and offered standard treatment with, adjuvant therapy. Follow-up is standardised to provide accurate data on recurrence and survival and more frequent examinations and investigations are performed if clinically indicated.

Frequency of Follow-up:

The minimum number of follow-up evaluations is as follows:

* every 3 months for the lst year.
* every 6 months for the 2nd and 3rd years.
* annually for the 4th and 5th years.

Test Schedule:

The minimal requirements for follow-up investigations are as follows:

* History and examination with a specific check for tumour wound recurrence.
* Colon evaluation including colonoscopy or sigmoidoscopy plus barium enema.
* Annual examination if positive for neoplasia (earlier if preoperative proximal examination is incomplete for technical reasons); examination every 3 years if negative.
* haemoglobin and white cell count
* creatinine, SGOT, alkaline phosphatase, total bilirubin, CEA
* Chest X-ray
* Abdominal CT scan or liver ultrasound annually for 5 years.
* Quality of Life and Complications documentation postoperatively at 2 days, 2 weeks, 2 months and 18 months.

SIGNIFICANCE AND OUTCOMES

The study will determine the efficacy and safety of laparoscopic assisted resection of colonic adenocarcinoma. It will also answer questions of cost effectiveness and quality of life improvement. It will determine if port site recurrence is a real issue in this type of surgery.

The study will also give valuable data about the outcomes of patients undergoing laparotomy in regard to current length of hospital stay, effectiveness of post-operative analgesia, in hospital complications and transfusion requirements.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a single adenocarcinoma of the ascending, descending, or sigmoid colon
* 18 years of age or older
* Able to give informed consent
* Must be able to participate in follow-up examinations
* Must not have prohibitive scars or adhesions from previous abdominal surgery

Exclusion Criteria:

* Advanced local disease, defined as >8cm in diameter or extensive infiltration
* Any previous or current malignant tumour with the previous 5 years (except superficial squamous or basal cell skin carcinoma or in situ cervical cancer)
* ASA 4
* ASA 5
* Associated gastrointestinal disease
* Dukes D disease
* Emergency presentation
* Massive bleeding
* Morbid obesity
* Pregnancy
* Rectal cancer
* Transverse colon cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 1998-01; Study Completion 2010-03

PRIMARY OUTCOMES:
Disease-free interval
Three-year survival
Five-year survival

SECONDARY OUTCOMES:
30-day mortality
Postoperative pain
Paralytic ileus
Early morbidity
Late morbidity
Recovery
Transfusion requirement
Cost effectiveness
Quality of Life outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Hewett, MBBS, FRACS, Study Director — The Queen Elizabeth Hospital; Andrew RL Stevenson, MBBS, FRACS, Principal Investigator — Royal Brisbane Hospital; Michael J Solomon, FRACS, MSc, Principal Investigator — Royal Prince Alfred Medical Centre
Locations (20):
- Australia (18):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Hospital, Concord, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Royal North Shore Hospital & Community Health Service, St Leonards, New South Wales
  - Wesley Hospital, Auchenflower, Queensland
  - Royal Brisbane Hospital, Brisbane, Queensland
  - Holy Spirit Northside Private Hospital, Chermside, Queensland
  - North West Brisbane Private Hospital, Everton Park, Queensland
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Lyell McEwin Health Service, Elizabeth Vale, South Australia
  - Calvary Health Care Adelaide Inc., North Adelaide, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Ballarat Base Hospital, Ballarat, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Western Health, Footscray, Victoria
  - Cabrini Institute, Malvern, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
- New Zealand (2):
  - Auckland Hospital, Auckland
  - Christchurch Hospital, Christchurch

REFERENCES:
- [Derived] Bagshaw PF, Allardyce RA, Frampton CM, Frizelle FA, Hewett PJ, McMurrick PJ, Rieger NA, Smith JS, Solomon MJ, Stevenson AR; Australasian Laparoscopic Colon Cancer Study Group. Long-term outcomes of the australasian randomized clinical trial comparing laparoscopic and conventional open surgical treatments for colon cancer: the Australasian Laparoscopic Colon Cancer Study trial. Ann Surg. 2012 Dec;256(6):915-9. doi: 10.1097/SLA.0b013e3182765ff8. PMID 23154392
- [Derived] Allardyce RA, Bagshaw PF, Frampton CM, Frizelle FA, Hewett PJ, Rieger NA, Smith JS, Solomon MJ, Stevenson AR; Australasian Laparoscopic Colon Cancer Study Group. Australasian Laparoscopic Colon Cancer Study shows that elderly patients may benefit from lower postoperative complication rates following laparoscopic versus open resection. Br J Surg. 2010 Jan;97(1):86-91. doi: 10.1002/bjs.6785. PMID 19937975
- [Derived] Hewett PJ, Allardyce RA, Bagshaw PF, Frampton CM, Frizelle FA, Rieger NA, Smith JS, Solomon MJ, Stephens JH, Stevenson AR. Short-term outcomes of the Australasian randomized clinical study comparing laparoscopic and conventional open surgical treatments for colon cancer: the ALCCaS trial. Ann Surg. 2008 Nov;248(5):728-38. doi: 10.1097/SLA.0b013e31818b7595. PMID 18948799